CLINICAL TRIAL: NCT00557219
Title: Influence of Fenoldopam and Ketanserin on Function and Kidney Injury Parameters in Patients With Increased Risk of Acute Kidney Failure After Cardiac Surgery
Brief Title: Fenoldopam and Ketanserin for Acute Kidney Failure Prevention After Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Main cooperator finished cooperation
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Maciej M. Kowalik, Dr., Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AMG-NKEBN/225/2007
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Acute Renal Failure
Keywords: cardiac surgery; fenoldopam; ketanserin; renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Fenoldopam; Ketanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Control group receiving placebo
  Interventions: Drug: placebo
- Ketanserin (Experimental): patients receiving ketanserin infusion
  Interventions: Drug: ketanserin (Sufrexal)
- Fenoldopam (Experimental): patients receiving fenoldopam infusion
  Interventions: Drug: fenoldopam (Corlopam)

INTERVENTIONS:
Drug: fenoldopam (Corlopam) — continuous intravenous infusion of 0.3 μg/kg/min fenoldopam for 24 hours
  Arms: Fenoldopam
Drug: placebo — continuous intravenous infusion of 2 mL/hour of 0.9% natrium chloride solution for 24 hours
  Arms: Placebo
Drug: ketanserin (Sufrexal) — continuous intravenous infusion 0.1 mg/kg/hour ketanserin for 24 hours
  Arms: Ketanserin

SUMMARY:
The purpose of the study is to compare the effect of fenoldopam and ketanserin on kidney function preservation in patients at high risk for renal failure after cardiac surgery. Acute, oliguric renal failure develops in up to 2% of patients undergoing cardiac surgery. Some of them require renal replacement therapy and despite that mortality in this group exceeds 30-60%. The investigators await that the use of fenoldopam and/or ketanserin may decrease the rate of severe renal failure.

DETAILED DESCRIPTION:
Informed, signed consent will be obtained from the patient before surgery. In patients with acute consciousness disorders, the consent will be obtained from a legal representative and confirmed by the local court - accordingly to Polish legacy.

Patients willing to participate into the study and fulfilling at least one of two inclusion criteria will be randomly assigned to one of the three study groups. The treatment will be applied for 24 hours.

Intention to treat analysis will include comparison for differences of continuous, homogeneous distributed data with use of parametric tests, parametric or inhomogeneous distributed data - with use of nonparametric tests. The treatment effect will be assessed by comparison of the odds ratios for primary and secondary outcomes between the groups.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery
* at least one risk factor for acute renal failure:

  1. oliguria < 0.5 ml/kg/hour for over 3 hours despite adequate blood volume and furosemide intravenously
  2. at least 60 mg furosemide/12 hours iv to maintain diuresis > 1 ml/kg/hour

Exclusion Criteria:

* refused or none consent
* chronic renal failure with chronic renal replacement therapy
* chronic increase of serum creatinine > 2 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cystatin C and NGAL in serum | after 24 and 48 hours from treatment start

SECONDARY OUTCOMES:
β2microglobulin in urine | after 24, 48 and 72 hours of treatment
creatinine increase in serum | after 24, 48 and 72 hours of treatment
frequency of renal replacement therapy | 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Klajbor, MD, Principal Investigator — Dept. of Cardiac Anesthesiology, Medical University of Gdańsk; Romuald Lango, MD, PhD, Study Director — Dept. of Cardiac Anesthesiology, Medical University of Gdańsk
Locations (1):
- Department of Cardiac Anesthesiology, Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request IPD can be made available to other researcher.

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014
- See also: home page of the Dept. of Cardiac Anesthesiology, MUG — http://www.informator.gumed.edu.pl/327